CLINICAL TRIAL: NCT03764228
Title: Single Arm Clinical Study of Human Amniotic Epithelial Cells in Preventing Acute Graft-versus-host Disease After Hematopoietic Stem Cell Transplantation
Brief Title: Human Amniotic Epithelial Cells Prevent Acute Graft-versus-host Disease After Hematopoietic Stem Cell Transplantation
Acronym: hAECs-GVHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Director of the Hematology Department, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018PHD006-01
Record Dates: First submitted 2018-11-29; First posted 2018-12-05 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Acute-graft-versus-host Disease
Keywords: human amniotic epithelial cells(hAECs); Acute-graft-versus-host disease（aGVHD）

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hAECs (Experimental): Infusion of hAECs at the day before HSCT and 7th days after HSCT. The dose is 1×10^6, 2×10^6, 5×10^6 cell/kg, successively.
  Interventions: Biological: hAECs

INTERVENTIONS:
Biological: hAECs — Human amniotic epithelial cells（hAECs）

SUMMARY:
This is a Single arm clinical study evaluating the safety and efficacy of hAECs in preventing aGVHD after HSCT.

DETAILED DESCRIPTION:
A dose escalation study evaluating the safety and efficacy of human amniotic epithelial cells( hAECs) in preventing acute graft-versus-host(aGVHD) disease after hematopoietic stem cell transplantation(HSCT). The doses were 1×10^6、2×10^6、5×^6 cell/kg, successively.

ELIGIBILITY:
Inclusion Criteria:

* Standard risk GVHD patients with hematological malignancies;
* High risk GVHD patients with hematological malignancies: haplotype hematopoietic stem cell transplantation patients, donor is female or more than 30 years old;
* Well informed about this study and signed a consent form before the trial;
* Left ventricular ejection fraction (LVEF) ≧ 50%, no evidence of pericardial effusion;
* No evidence of lung infection by X-rays examination;
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1, Hematopoietic cell transplantation - specific comorbidity index (HCT-CI) of 0, 1, 2;
* Normal liver and kidney function;

Exclusion Criteria:

* Reduce pretreatment dose or secondary transplantation;
* participate other clinical trials within 2 months before this study;
* Female, 1) pregnant/nursing period, or 2) have a pregnancy plan during the study period, or 3) have fertility and cannot take effective contraception;
* History of severe allergic disease or is allergic to one or more drugs;
* Patients who are considered unsuitable for the study by the investigator.

Ages: 8 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events | 1 year
  Safety of HSCT combined with hAECs infusion;

SECONDARY OUTCOMES:
GVHD | 1 year
  Occurrence of Graft-versus-host disease after hAECs infusion

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Principal Investigator — Peking University People's Hospital
Locations (2):
- China (2):
  - Peking University Institute of Hematology, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality

REFERENCES:
- [Derived] Yang PJ, Zhao XY, Kou YH, Liu J, Ren XY, Zhang YY, Wang ZD, Ge Z, Yuan WX, Qiu C, Tan B, Liu Q, Shi YN, Jiang YQ, Qiu C, Guo LH, Li JY, Huang XJ, Yu LY. Human amniotic epithelial stem cell is a cell therapy candidate for preventing acute graft-versus-host disease. Acta Pharmacol Sin. 2024 Nov;45(11):2339-2353. doi: 10.1038/s41401-024-01283-y. Epub 2024 May 27. PMID 38802569